CLINICAL TRIAL: NCT02136004
Title: The Closer Trial: A Multi-center, Prospective, Single Arm Trial to Evaluate the Safety and Efficacy of the Rex Medical Closer Vascular Sealing System (VSS) for the Management of the Femoral Arteriotomy After Percutaneous Endovascular Procedures
Brief Title: The Closer Trial: A Safety and Efficacy Study of the Rex Medical Vascular Sealing System
Acronym: Closer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rex Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REX-US-2027-001
Record Dates: First submitted 2014-05-07; First posted 2014-05-12 (Estimated); Results first posted 2016-12-29 (Estimated); Last update posted 2017-10-27 (Actual); Status verified 2017-09

CONDITIONS: Surgical Wound
Keywords: arteriotomy; vessel closure; femoral access site
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Closer VSS (Experimental): Rex Medical Closer Vascular Sealing System to close femoral arteriotomy
  Interventions: Device: Closer VSS

INTERVENTIONS:
Device: Closer VSS — At the end of a percutaneous endovascular procedure, the femoral arterial access site is closed with the Closer device to achieve arterial hemostasis.
  Other Names: Rex Medical Closer TM Vascular Sealing System (VSS)

SUMMARY:
The objective of this trial is to demonstrate the safety and effectiveness of the Rex Medical Closer Vascular Sealing System in sealing femoral arterial access sites.

DETAILED DESCRIPTION:
The objective of the trial is to demonstrate the safety and effectiveness of the Rex Medical Closer Vascular Sealing System (VSS) in sealing femoral arterial access sites and providing reduced times to hemostasis (TTH) compared with performance goals at the completion of diagnostic or interventional procedures performed through 5, 6 or 7 Fr procedural sheaths. This study will be considered a success (from a statistical perspective) if it meets both the Closer VSS superiority goal for the primary effectiveness analysis and the Closer VSS performance goal for the primary safety analysis.

ELIGIBILITY:
Inclusion Criteria:

Pre-Op Inclusion Criteria:

1 - Acceptable candidates for an elective, non-emergent diagnostic or interventional endovascular procedure via the common femoral artery using a 5, 6, or 7 Fr introducer sheath.

-

Exclusion Criteria:

Pre-Operative Exclusion Criteria:

1. - Significant bleeding diatheses or coagulopathy
2. - Planned endovascular or surgical procedures within next 30 days
3. - Planned ipsilateral femoral arteriotomy within next 90 days
4. - Arteriotomy in ipsilateral groin within the past 30 days with any residual hematoma, significant bruising or vascular complication
5. - Previous vessel closure device used in ipsilateral groin within the past 90 days
6. - Previous vascular surgery or repair in the vicinity of the target access site
7. - Severe peripheral vascular disease in the ipsilateral limb requiring surgical or endovascular treatment within the pervious 30 days or next 30 days
8. - Existing nerve damage in ipsilateral limb
9. - Extreme morbid obesity (BMI > 4 kg/m2)

   Intra-operative Exclusion Criteria:
10. - Use of a procedural sheath that is < 5 Fr or > 7 Fr
11. - Difficult insertion of procedural sheath or needle stick problems at the onset of the procedure
12. - Placement of an ipsilateral venous sheath for procedure
13. - Procedural sheath placement either through the superficial femoral artery and into the profunda femoris artery, or placement at or distal to bifurcation of the superficial femoral artery and the profunda femoris artery
14. - In subjects receiving unfractionated heparin, an ACT > 350 seconds, or > 250 seconds in the presence of a GP IIb/IIIa inhibitor
15. - Procedures or existing medical conditions that may extend index hospitalization beyond 24 hours post-procedure
16. - Systemic hypertension (SBP > 180 mmHg) or hypotension (SBP < 90 mmHg) just prior to enrollment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shing-Chiu Wong, MD, Principal Investigator — New York Presbyterian Hospital
Locations (12):
- United States (12):
  - UC Davis Medical Center, Sacramento, California
  - Colorado Neurological Institute, Englewood, Colorado
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Lafayette General Medical Center/Cardiovascular Institute of the South, Lafayette, Louisiana
  - New York Presbyterian Hospital, New York, New York
  - North Ohio Research, Elyria, Ohio
  - Oklahoma Heart Institute, Tulsa, Oklahoma
  - Oregon Health & Science University, Portland, Oregon
  - Geisinger Health Center, Danville, Pennsylvania
  - Geisinger Health Center, Wilkes-Barre, Pennsylvania
  - Pinnacle Health, Wormleysburg, Pennsylvania
  - Heart Hospital of Austin, Austin, Texas

IPD SHARING:
Plan to Share IPD: Yes
After multi-center manuscript is published.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Closer VSS
Started | 220 (Enrollment commenced on May 20, 2014 and the last subject completed follow-up on February 28, 2015)
Completed | 219
Not Completed | 1

BASELINE CHARACTERISTICS:
Groups:
- Closer VSS - Diagnostic Cohort: Rex Medical Closer Vascular Sealing System to close femoral arteriotomies in diagnostic endovascular cases.
  Closer VSS: At the end of a percutaneous diagnostic endovascular procedure, the femoral arterial access site is closed with the Closer device to achieve arterial hemostasis.
- Closer VSS - Interventional Cohort: Rex Medical Closer Vascular Sealing System to close femoral arteriotomies in interventional endovascular cases.
  Closer VSS: At the end of a percutaneous interventional endovascular procedure, the femoral arterial access site is closed with the Closer device to achieve arterial hemostasis.
- Total: Total of all reporting groups
Arm/Group | Closer VSS - Diagnostic Cohort | Closer VSS - Interventional Cohort | Total
Number analyzed (Participants) | 111 | 109 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.2 (10.3) | 64.7 (8.7) | 63.9 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 25 | 70
  Male | 66 | 84 | 150

OUTCOME MEASURES:

1. Primary Outcome: Time to Hemostasis
Description: Primary effectiveness endpoint - elapsed time between the Closer VSS delivery system removal and first observed and confirmed arterial hemostasis
Time Frame: procedural, usually within 15 minutes of enrollment
Population: All subjects enrolled
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | Closer VSS
Number analyzed (Participants) | 220
minutes | 1.78 [0.74 to 2.82]

2. Primary Outcome: Rate of Combined Major Access Site Closure-related Complications
Description: Primary safety endpoint - rate of combined major access site closure-related complications
Time Frame: Through 30 days +/- 7 days
Population: All subjects enrolled
Measure: Number; unit: complications
Arm/Group | Closer VSS
Number analyzed (Participants) | 220
complications | 0

3. Secondary Outcome: Time to Ambulation
Description: Secondary efficacy endpoint - elapsed time between the Closer VSS delivery system removal and when subject stands and walks 20 feet without evidence of arterial re-bleeding from the access site
Time Frame: prior to hospital discharge, usually within 24 hours
Population: All subjects enrolled
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Closer VSS
Number analyzed (Participants) | 220
hours | 2.50 [2.36 to 2.64]

4. Secondary Outcome: Time to Discharge Eligibility
Description: Secondary efficacy endpoint - elapsed time between Closer VSS delivery system removal and when subject's access site is assessed to be hemodynamically stable, as determined by the investigator or his/her designee(s)
Time Frame: prior to hospital discharge, usually within 24 hours
Population: All subjects enrolled
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Closer VSS
Number analyzed (Participants) | 220
hours | 2.83 [2.62 to 3.03]

5. Secondary Outcome: Time to Hospital Discharge
Description: Secondary efficacy endpoint - elapsed time between Closer VSS delivery system removal and when subject is actually physically discharged from the hospital ward
Time Frame: through hospital discharge, usually within 24 hours
Population: All subjects enrolled
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Closer VSS
Number analyzed (Participants) | 220
hours | 13.12 [10.93 to 15.32]

6. Secondary Outcome: Device Success
Description: Secondary efficacy endpoint - the ability to deploy the system, deliver the implant, and achieve arterial hemostasis with the Closer VSS alone or with post-hemostasis adjunctive compression
Time Frame: procedural, usually within 15 minutes of enrollment
Population: All subjects enrolled
Measure: Count of Participants; unit: Participants
Arm/Group | Closer VSS
Number analyzed (Participants) | 220
Participants | 216

7. Secondary Outcome: Rate of Combined Minor Access Site Closure-related Complications
Description: Secondary safety endpoint - rate of combined minor access site closure-related complications
Time Frame: through 30 +/- 7 days
Population: All subjects enrolled
Measure: Number; unit: complications
Arm/Group | Closer VSS
Number analyzed (Participants) | 220
complications | 3

8. Secondary Outcome: Procedure Success
Description: Secondary efficacy endpoint - attainment of final arterial hemostasis using any method and freedom from major access site closure-related complications through 30 days
Time Frame: through 30 days +/- 7 days
Population: All subjects enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Closer VSS
Number analyzed (Participants) | 219
Participants | 219

ADVERSE EVENTS:
Arm/Group | Closer VSS
Serious Adverse Events (participants affected / at risk) | 0/220
Other Adverse Events (participants affected / at risk) | 12/220
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closer VSS (N=220)
Serious device-related adverse events, excluding endpoint events (Vascular disorders) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Closer VSS (N=220)
Non-serious access site bleeding (Vascular disorders) | 12 (12)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No